CLINICAL TRIAL: NCT03213223
Title: Retention-in-care of Women in the Elimination of Mother-to-child Transmission of HIV (eMTCT) Option B Plus Program in Mashonaland East, Zimbabwe: a Mixed Method Study
Brief Title: Retention of Women in the PMTCT (Prevention of Mother-to-child Transmission of HIV)
Status: Completed | Type: Observational
Sponsor: University of Zimbabwe (Other)
Collaborators: NORHED (Unknown)
Responsible Party: Principal Investigator, Augustine Ndaimani, (Lecturer, Faculty of Medicine, Principal Investigator, DPhil Student)., University of Zimbabwe
Other Study IDs: A2087
Record Dates: First submitted 2017-06-30; First posted 2017-07-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Prevention of Mother-to-child Transmission of HIV
Keywords: retention; attrition; PMTCT; elimination of mother to child transmission of HIV
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
EXECUTIVE SUMMARY RESEARCH QUESTION TO BE ADDRESSED BY THIS PROPOSAL What are the factors associated with retention-in-care of women enrolled in the eMTCT Option B+ program at eMTCT (elimination of mother-to-child transmission of HIV) sites with high retention-in-care compared to eMTCT sites with low retention in care? Hypotheses Null hypothesis H0: The attributable rate of low retention-in-care of women in the eMTCT program at eMTCT sites equals zero.

Alternative hypothesis HA: The attributable risk of low retention-in-care of women in the eMTCT program at eMTCT sites is not equal to zero.

RATIONALE FOR RESEARCH There is poor retention of women along the PMTCT (prevention of mother to child transmission of HIV) cascade. Retention in eMTCT refers to documented regular participation of the pregnant woman, confirmed HIV positive, together with her child or children not yet confirmed as HIV-positive, in all prescribed activities aimed at preventing transmission of HIV from her to the child, and scheduled or unscheduled HIV-care related visits, measured during or at the end of care. It results in uninterrupted supply of ART (antiretroviral therapy). Retention in PMTCT ranges between 10.6% and 76.5% in other countries. In Zimbabwe it was found to drop from 83% at second pick up of antiretroviral drugs to 45% at fourth pick up of antiretroviral drugs. Poor retention in PMTCT leads to poor health outcomes in the mother and the baby. These include increased viral load, reduced CD4 count, reduced adherence to ART, emergency of drug resistant HIV strains, reduced quality of life, increased frequency of opportunistic infections, increased all-cause hospitalizations and death of women and children. HIV infection contributes to between 6 and 20% of maternal deaths. On the other hand, about 14% of all new infections are due to MTCT (mother to child transmission of HIV).

Retention in care is better at some clinics and hospitals. The purpose of the study will be to determine the factors associated with retention-in-care of women enrolled in the eMTCT Option B+ program at eMTCT sites.

The following objectives will be addressed in the study:

1. To assess the PMTCT Option B Plus program at selected eMTCT sites.
2. To determine the prevalence of retention among women enrolled in the eMTCT Option B+ program at selected eMTCT sites.
3. To determine the incidence of attrition among women enrolled in the eMTCT Option B+ program at selected eMTCT sites.
4. To identify factors associated with variability in levels of retention-in-care of women in the eMTCT Option B+ program at selected eMTCT sites.
5. To explore the barriers and facilitators of retention among women enrolled in the eMTCT Option B+ program.

METHODS The study is being done through a nested, embedded, mixed methods study with priority given to a prospective cohort methodology. The supplementary design is a simple descriptive qualitative design carried out through focus group discussions. A mixed methods design caters for the weaknesses in either a qualitative or a quantitative design. Hence, it is ideal in study of complex human issues such as retention in the PMTCT Option B Plus program.

In the study, 462 pregnant women enrolled for PMTCT Option B Plus will be followed up for 12 months in an open cohort. The sample size was calculated using Stata software based on a power of 0.8, a margin of error of 0.05, a design effect of 1.1 and a retention rate of 0.45. Six randomly selected eMTCT sites in Mashonaland East Province were chosen for the study. Retention rate at the sites since 2013 will be calculated. Three sites with lower retention will be considered as the exposure sites. The other 3 sites will be the unexposed sites. Option B Plus, a recently introduced and recommended PMTCT option, was meant to benefit pregnant women, in addition to their children and sexual partners. Hence, the involvement of women as participants. Four focus group discussions will also be done, with nursing mothers to ascertain the barriers and facilitators of retention in PMTCT Option B plus. Included in the study will be HIV positive pregnant and nursing women coming for PMTCT Option B Plus. Women who can communicate in English or Shona and are without psychiatric conditions will also be included. Emancipated minors, below 18 years of age will also be included. Excluded from the study will be women enrolled in PMTCT Options A or B, women with psychiatric conditions or those who are too ill to participate. The study was approved by The Medical Research Council of Zimbabwe. Signed voluntary consent is sought from participants. Data is being collected through questionnaires and audio-taped focus group discussions. Follow-up data will also be extracted from eMTCT registers at respective eMTCT sites. Data is kept in locked cabinets only accessible to the principal investigator and the supervisors.

ELIGIBILITY:
Inclusion Criteria:

* women 15-49 years. On PMTCT tes and treat strategy or Option B+

Exclusion Criteria:

* mentally unstable women or not enrolled at the study sites for PMTCT. Women enrolled in Option B Censoring - after a miscarriage, still birth, on leaving the PMTCT program and at the end of the study

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant or breastfeeding women in the PMTCT program
Study Population: The target population in the study will consist of women who are enrolled in eMTCT Option B+ program. The accessible population will be women enrolled and coming for PMTCT services at eMTCT sites in Mashonaland East Province.
Sampling Method: Probability Sample
Enrollment: 468 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Retention in care based on record review and follow up data | One follow-up per 3-month period, up to 12 months
  Missed visit count (number of missed visits), Dichotomous missed visit (more than one missed visit), Visit adherence (number of kept visits divided by the total number of scheduled visits), Four month constancy (the number of four month intervals in which the individual came for PMTCT at least once), 6-month gap (no visit in a 6-month period), HRSA HAB (Health Resources and Services administration HIV-AIDS Bureau) [2 kept visits separated by at least 90 days in a year)
Attrition from PMTCT (determined through survival analysis based on Cox proportional hazards regression) | One follow-up per 3-month period, up to 12 months
  Death or loss to follow - up from PMTCT

SECONDARY OUTCOMES:
Barriers and enablers of retention (focus group discussions) | One focus group per week, up to 4 weeks, (total of four focus group discussions)
  Perceived barriers and facilitators of retention. Focus group discussions analysed through latent content analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Augustine Ndaimani, DPhil MD (Student), Principal Investigator — University of Zimbabwe
Locations (1):
- Mashonaland East Province (Mutoko Hospital, Murewa Hospital, Kunaka Hospital, Nharira Hospital, Chichu Clinic, Epworth Polyclinic), Marondera, Mashonaland East Province, Zimbabwe

IPD SHARING:
Plan to Share IPD: No